CLINICAL TRIAL: NCT03906240
Title: Using Moral Elevation to Improve Functioning in Veterans With PTSD and Moral Injury: A Pilot Study of a Web-Based Intervention
Brief Title: Pilot Study Testing a Web-Based Moral Elevation Intervention for Veterans With PTSD and Moral Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3035-P
Record Dates: First submitted 2019-03-27; First posted 2019-04-08 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Posttraumatic Stress Disorder; Moral Injury
Keywords: Web-Based Intervention; Pilot Study; Moral Elevation; Veterans; PTSD; Moral Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either an intervention condition or no-treatment condition. The intervention condition is accessed through an online portal and includes the moral elevation intervention with intervention content and session goals to facilitate social engagement. The no-treatment condition includes accessing the same online portal, but without any intervention content and is limited to repeated self-report measures for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No intervention (No Intervention): Veterans will access the online portal and complete session measures, but will not be presented with any intervention content (i.e., videos, journaling exercise, and goal setting exercise)
- Moral Elevation Intervention (Experimental): Moral Elevation Intervention (described in intervention section).
  Interventions: Behavioral: Moral Elevation intervention

INTERVENTIONS:
Behavioral: Moral Elevation intervention — The intervention will be administered twice per week for 8 sessions total. The intervention will include two types of moral elevation exercises related to witnessing virtuous behavior and subsequently setting session goals aimed to facilitate social engagement.
  Arms: Moral Elevation Intervention

SUMMARY:
Given the prevalence of posttraumatic stress disorder (PTSD) and moral injury in combat Veterans and the limitations to current treatments, novel approaches are needed to target both PTSD and moral injury and directly impact psychosocial growth and functional recovery. One potential way to address this critical need is through moral elevation-a positive emotional state described as feeling uplifted and inspired by others' virtuous actions. This study will pilot a web-based moral elevation intervention with Operations Enduring Freedom, Iraqi Freedom, and New Dawn Veterans who experienced a morally injurious event and with a PTSD diagnosis. If Veterans are willing and able to complete an online moral elevation intervention and it has beneficial effects, then moral elevation could be feasibly utilized as a tool to reverse the negative effects of trauma and facilitate recovery. Data from this study will be used to develop larger clinical trials to test if this intervention significantly improves PTSD symptoms and moral injury distress and enhances social functioning.

DETAILED DESCRIPTION:
The goal of this proposed study is to conduct a pilot trial of a web-based moral elevation intervention to determine if such an intervention is a feasible and acceptable therapeutic approach for Operations Enduring Freedom, Iraqi Freedom, and New Dawn Veterans with distress related to posttraumatic stress disorder (PTSD) and moral injury (MI). This study will also assess the feasibility of randomization, retention, and completion of a no-treatment condition (i.e., comparison group) in preparation for future randomized controlled trials (RCTs). The sample will include 24 Veterans (12 per group). The online intervention consists of two exercises per week for one month, totaling eight sessions. Sessions will include watching validated videos that elicit moral elevation and recalling moments when one experienced moral elevation in daily life, paired with journaling about one's reactions to witnessed virtuous behavior. Participants in the intervention condition will also be presented with a brief goal to be completed prior to the next session to facilitate greater social engagement. Participants randomized to the no-treatment condition will access the same online portal twice per week, but will not be exposed to any intervention components. All participants will complete brief self-report measures at each online session. All participants will also complete self-report measures at baseline and 1-month follow-up that will assess PTSD symptoms, MI distress, prosocial behavior, and quality of social relationships. At the follow-up assessment, participants randomized to the intervention condition will complete an individual qualitative interview with a member of the study team to assess acceptability and satisfaction with the intervention and proposed methodology, which will be coded and analyzed to inform future clinical trials. To supplement self-report measures, all participants will invite a significant other (e.g., spouse, close friend) to complete measures based on observations of the Veteran's behavior and social functioning at baseline and 1-month follow-up. Feasibility of recruitment, retention, and completion of the intervention will be analyzed by tracking the number of participants retained at each stage of the study, as well as the number of sessions completed in the intervention. Results from this study will be used to develop an RCT with a larger sample size to determine the efficacy of a moral elevation intervention and assess whether this novel approach leads to unique beneficial outcomes regarding PTSD and moral injury distress.

ELIGIBILITY:
Inclusion Criteria:

Veteran Participant Inclusion Criteria:

* 18 years of age
* OEF/OIF/OND Veteran enrolled in CTVHCS
* English-speaking and able to provide written informed consent
* Internet access for web-based sessions and measures
* Current PTSD diagnosis based on medical chart review or screen positively for a probable diagnosis based on empirically-validated cutoffs on the PTSD Checklist for DSM-5
* Screen positively for experiencing 1 morally injurious event and endorse some distress (>4 on any item) related to that event based on the Moral Injury Events Scale (MIES)
* Willing to complete study procedures and identify an SO who will complete observational measures
* Willing to be randomized

Significant Other Participant Inclusion Criteria:

* 18 years of age
* Designated as a Significant Other by the Veteran participant, and the Veteran participant has provided consent for the study team to contact that potential Significant Other
* English-speaking
* Internet access for web-based observational measures
* Interact with the Veteran >1 time per week
* Willing to complete study procedures

Exclusion Criteria:

Veteran Participant Exclusion Criteria:

* History of severe traumatic brain injury indicated by medical review and the Ohio State Traumatic Brain Injury Identification Method (OSU TBI-ID)
* Psychosis or current substance use disorder indicated by medical review and the Mini International Neuropsychiatric Interview (MINI)
* Current suicide risk based on the Beck Depression Inventory-II (BDI-II)

Significant Other Participant Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam P. McGuire, PhD, Principal Investigator — Central Texas Veterans Health Care System, Temple, TX
Locations (1):
- Central Texas Veterans Health Care System, Temple, TX, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Time Frame: 1 year after publication

REFERENCES:
- [Derived] McGuire AP, Rodenbaugh M, Howard BAN, Contractor AA. Response styles to positive affect during a positive psychology intervention for veterans with PTSD and moral injury: Preliminary results from a moral elevation intervention pilot trial. Psychol Trauma. 2025 Feb;17(2):457-465. doi: 10.1037/tra0001774. Epub 2024 Aug 29. PMID 39207432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among 87 participants who were eligible following the initial pre-screen (phone), 48 were determined to be eligible and randomized.
Groups:
- Moral Elevation Intervention: Moral Elevation Intervention (described in intervention section).
  Moral Elevation intervention: The intervention was administered twice per week for 8 sessions total. The intervention included two types of moral elevation exercises related to witnessing virtuous behavior and subsequently setting session goals aimed to facilitate social engagement.
- No Intervention: Veterans accessed the online portal and complete session measures, but were not be presented with any intervention content (i.e., videos, journaling exercise, and goal setting exercise)
Period: Overall Study
Arm/Group | Moral Elevation Intervention | No Intervention
Started | 24 | 24
Completed (Participants who completed greater than 4 out of 8 sessions were considered to have completed the intervention.) | 19 | 23
Not Completed | 5 | 1
Not completed — Failed to complete Session 1 (essential orientation), thus excluded from future sessions. | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Moral Elevation Intervention: Moral Elevation intervention: The intervention was administered twice per week for 8 sessions total. The intervention included two types of moral elevation exercises related to witnessing virtuous behavior and subsequently setting session goals aimed to facilitate social engagement.
- Total: Total of all reporting groups
Arm/Group | Moral Elevation Intervention | No Intervention | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.42 (6.45) | 45.38 (8.85) | 44.40 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 18 | 22 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 6 | 10 | 16
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 6 | 3 | 9
PTSD Symptoms [Mean (Standard Deviation); unit: score on a scale] — Posttraumatic Checklist for DSM-5, total score ranging from 0 to 80. Higher scores indicate greater symptom severity. (PCL-5; Weathers et al., 2013).
  score on a scale | 61.93 (8.74) | 53.70 (11.46) | 57.82 (10.90)
Moral Injury Event Exposure [Mean (Standard Deviation); unit: score on a scale] — Moral Injury Events Scale, total range is 11 to 66, with higher scores reflecting greater moral injury. (MIES; Nash et al., 2013).
  score on a scale | 35.38 (7.15) | 31.58 (8.50) | 33.48 (8.00)
Moral Injury-Related Distress [Mean (Standard Deviation); unit: score on a scale] — Expression of Moral Injury Scale, total score ranging from 17 to 85. Higher scores indicate greater moral injury-related distress. (EMIS; Currier et al., 2018).
  score on a scale | 55.39 (16.65) | 57.79 (12.95) | 56.62 (14.77)
Quality of Life [Mean (Standard Deviation); unit: score on a scale] — The World Health Organization Quality of Life includes 4 subscales: Physical Domain (7 items), Psychological Domain (6 items), Social Domain (3 items), and Environment Domain (8 items). Subscales scores are computed by summing all items for each subscale, then all scores are transformed to a range of 0-100. A higher score signifies higher or better quality of life. (WHOQOL-BREF Group et al., 1998).
  score on a scale
    Physical Domain | 39.75 (12.80) | 39.58 (19.92) | 39.67 (16.64)
    Psychological Domain | 37.05 (14.32) | 35.94 (19.96) | 36.48 (17.25)
    Social Domain | 43.75 (25.49) | 41.67 (20.57) | 42.64 (22.73)
    Environment Domain | 58.45 (19.80) | 57.45 (20.32) | 57.94 (19.86)
Prosocial Behavior [Mean (Standard Deviation); unit: score on a scale] — Prosocialness Scale, total score ranging from 16 to 80. Higher scores indicate greater prosocial behavior. (PS; Caprara et al., 2005).
  score on a scale | 53.43 (12.31) | 51.71 (14.24) | 52.55 (13.22)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Evaluation Inventory-Short Form (TEI-SF)
Description: The TEI-SF is a 9-item self-report measure that assessed acceptability of the moral elevation intervention and its procedure. Items were scored from 1 to 5, with higher scores indicating greater acceptability. To assess the acceptability of the treatment in this study, we calculated descriptive statistics to determine the average score for each item across the intervention condition. The mid-point item score for this measure (range = 1-5, mid-point = 3) was used as an indicator for adequate acceptability (e.g., average/medium levels of acceptability, or higher). Thus, item scores that were greater than 3 are interpreted as supporting medium to high perceived acceptability of the intervention.
Time Frame: Follow-up assessment within 1 week of study completion.
Population: Among the 24 participants randomized to the treatment condition, 16 completed the post-treatment survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moral Elevation Intervention
Number analyzed (Participants) | 16
units on a scale
  1. Acceptable way of dealing with problems related to PTSD and moral injury. | 3.62 (1.01)
  2. Willing to use this procedure again. | 4.00 (0.95)
  3. Like the procedures used in this intervention. | 3.94 (0.91)
  4. Believe the intervention is likely to be effective. | 3.69 (0.93)
  5. Believe others would experience discomfort during this intervention. | 2.75 (0.92)
  6. Believe intervention is likely to result in permanent improvement. | 3.25 (0.67)
  7. Overall, I have a positive reaction to this intervention. | 3.94 (0.84)

2. Primary Outcome: Exercise-Specific Satisfaction Survey (ESSS)
Description: The ESSS is a 4-item self-report measure that assessed acceptability of and satisfaction with the moral elevation exercises within the intervention condition. Items are scored from 0 to 8 with higher scores indicate greater perceived helpfulness and satisfaction with moral elevation exercises. To assess the satisfaction of the session components, we calculated descriptive statistics to determine the average score for each item across all 8 sessions (e.g., average score of item #1 for 8 repeated measurements across 8 sessions). The mid-point item score for this measure (range = 0-8, mid-point = 4) was used as an indicator for adequate satisfaction. Thus, item scores that were greater than 4 are interpreted as supporting medium to high perceived satisfaction of the intervention.
Time Frame: Repeated measure administered during online sessions 1-8 (every Monday & Thursday for 4 weeks of study participation). Participant scores for each item were averaged across all 8 sessions/measurements.
Population: This analysis of descriptive statistics across 8 sessions includes all participants who completed more than 4 sessions. Note: 3 of these participants completed the session surveys, but did not complete the final follow-up survey; thus, the discrepancy in sample sizes for outcome data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moral Elevation Intervention
Number analyzed (Participants) | 19
units on a scale
  1. Rate how helpful this session was to you. | 4.95 (2.37)
  2. Rate how much you benefitted from this session's exercise. | 4.64 (2.69)
  3. Rate how helpful the goal assignment was to you. | 5.11 (2.59)
  4. Rate how much you were fully engaged with the material for this session. | 6.22 (1.87)

3. Secondary Outcome: Elevation Scale (ES)
Description: The ES is a 12-item self-report measure of the degree to which state-level moral elevation is experienced. Items are scored from 0 to 4. Scores on 12 items were averaged to create a mean item score ranging from 0 to 4. Higher total scores indicate higher levels of state moral elevation. To assess the level of elevation elicited in sessions, we calculated descriptive statistics to determine the average elevation score for 8 repeated measurements across 8 sessions. The mid-point item score for this measure (range = 0-4, mid-point = 2) was used as an indicator for adequate elevation. Thus, an average elevation score that was greater than 2 is interpreted as supporting medium to high levels of elevation elicited in intervention sessions.
Time Frame: Repeated measure administered during online sessions 1-8 (every Monday & Thursday for 4 weeks of study participation). Participant scores were averaged across all 8 sessions/measurements.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moral Elevation Intervention
Number analyzed (Participants) | 19
units on a scale | 1.63 (1.12)

4. Other Pre Specified Outcome: Change From Baseline in Posttraumatic Checklist for DSM-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure that assessed PTSD symptom severity. Items were scored from 0 to 4 and summed to create a total score ranging from 0 to 80. Higher scores indicate greater symptom severity. Reported findings indicate changes in PCL-5 from baseline to follow-up across both conditions. Reported findings in the Outcome Measure Data Table represent PCL-5 scores at baseline and follow up assessments within each condition.
Time Frame: Administered at baseline and follow-up assessment within 1 week of study completion.
Population: Analysis includes all participants who were randomized to a condition and completed the follow-up survey.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Moral Elevation Intervention | No Intervention
Number analyzed (Participants) | 16 | 20
Scores on a Scale
  Baseline | 61.27 (8.54) | 52.34 (11.40)
  Follow-up | 43.56 (16.37) | 43.30 (17.05)
Statistical Analysis 1: Comparison: Moral Elevation Intervention; Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p < .001, t-test, 2 sided; t = 5.78; Cohen's d = 1.44, 95% CI 2-sided [1.00 to 2.49]
Statistical Analysis 2: Comparison: No Intervention; Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .002, t-test, 2 sided; t = 3.48; Cohen's d = 0.78, 95% CI 2-sided [0.35 to 1.38]

5. Other Pre Specified Outcome: Changes From Baseline in Expression of Moral Injury Scale-Military Version (EMIS-M)
Description: The EMIS-M is a 17-item self-report measure of expressions of distress related to a moral injury directed at both self and others. Items were scored from 1 to 5 and summed to create a total score ranging from 17 to 85. Higher scores indicate greater moral injury-related distress. Reported findings in the Outcome Measure Data Table represent EMIS-M scores at baseline and follow-up assessments within each condition.
Time Frame: Administered at baseline and follow-up assessment within 1 week of study completion.
Population: Analysis includes all participants who were randomized to a condition and completed the follow-up survey. For the intervention condition, 1 participant did not complete this survey at follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Moral Elevation Intervention | No Intervention
Number analyzed (Participants) | 15 | 20
Scores on a Scale
  Baseline | 53.93 (17.43) | 57.40 (13.29)
  Follow-up | 53.73 (17.65) | 53.75 (13.43)
Statistical Analysis 1: Comparison: Moral Elevation Intervention; Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .957, t-test, 2 sided; t = 0.06; Cohen's d = 0.01, 95% CI 2-sided [-0.45 to 0.91]
Statistical Analysis 2: Comparison: No Intervention; Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .033, t-test, 2 sided; t = 2.30; Cohen's d = 0.51, 95% CI 2-sided [0.08 to 1.25]

6. Other Pre Specified Outcome: Changes From Baseline in World Health Organization Quality of Life (WHOQOL-BREF)
Description: The WHOQOL-BREF is a 26-item self-report measure of overall quality of life with 4 domains (physical health, psychological health, social relationships, and environment) and was used to assess perceptions of psychological health and quality of social relationships. Subscales scores are computed by summing all items for each subscale, then all scores are transformed to a range of 0-100. A higher score signifies higher or better quality of life. Reported findings in the Outcome Measure Data Table represent the WHOQOL-BREF subscale scores at baseline and follow up assessments within each condition.
Time Frame: Administered at baseline and follow-up assessment within 1 week of study completion.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Moral Elevation Intervention | No Intervention
Number analyzed (Participants) | 15 | 20
Scores on a scale
  Physical Domain: Baseline | 39.05 (13.05) | 41.43 (21.03)
  Physical Domain: Follow-up | 47.62 (15.25) | 41.61 (17.96)
  Psychological Domain: Baseline | 40.97 (14.89) | 35.63 (19.14)
  Psychological Domain: Follow-up | 48.61 (18.34) | 37.92 (20.89)
  Social Domain: Baseline | 47.92 (27.55) | 43.42 (21.62)
  Social Domain: Follow-up | 54.86 (24.74) | 42.98 (21.56)
  Environmental Domain: Baseline | 59.83 (18.82) | 60.03 (18.99)
  Environmental Domain: Follow-up | 64.58 (20.48) | 59.69 (18.30)
Statistical Analysis 1: Comparison: Moral Elevation Intervention; Physical Domain: Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .015, t-test, 2 sided; t = 2.76; Cohen's d = 0.71, 95% CI 2-sided [0.32 to 1.31]
Statistical Analysis 2: Comparison: Moral Elevation Intervention; Psychological Domain: Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .012, t-test, 2 sided; t = 2.87; Cohen's d = 0.74, 95% CI 2-sided [0.26 to 1.55]
Statistical Analysis 3: Comparison: No Intervention; Physical Domain: Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .941, t-test, 2 sided; t = 0.08; Cohen's d = 0.02, 95% CI 2-sided [-0.43 to 0.55]
Statistical Analysis 4: Comparison: No Intervention; Psychological Domain: Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .270, t-test, 2 sided; t = 1.14; Cohen's d = 0.25, 95% CI 2-sided [-0.17 to 0.79]

7. Other Pre Specified Outcome: Changes From Baseline in Prosocialness Scale (PS) - Self-report
Description: The PS is a 16-item measure that was completed by Veterans (self-report) to assess their prosocial behaviors and tendencies to help others. Items were scored from 1 to 5 and summed to create a total score ranging from 16 to 80. Higher scores indicate greater prosocial behavior. Reported findings in the Outcome Measure Data Table represent PS scores at baseline and follow-up assessments within each condition.
Time Frame: Administered at baseline and follow-up assessment within 1 week of study completion.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Moral Elevation Intervention | No Intervention
Number analyzed (Participants) | 15 | 20
Scores on a Scale
  Baseline | 53.60 (12.79) | 52.95 (13.98)
  Follow-up | 52.33 (15.93) | 53.00 (13.40)
Statistical Analysis 1: Comparison: Moral Elevation Intervention; Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .768, t-test, 2 sided; t = 0.30; Cohen's d = 0.08, 95% CI 2-sided [-0.45 to 0.71]
Statistical Analysis 2: Comparison: No Intervention; Paired-samples t-test to conduct within-person comparison between baseline and follow-up; Test type: Superiority; p = .975, t-test, 2 sided; t = 0.05; Cohen's d = 0.01, 95% CI 2-sided [-0.53 to 0.42]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Moral Elevation Intervention | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
The main aim of this pilot trial was to test the feasibility and acceptability of the intervention. Therefore, statistical tests used for secondary/targeted outcomes should be interpreted with caution given the small sample size. Additionally, larger samples are needed to formally test between-group comparisons in change scores. Lastly, the state elevation measure did not perform optimally in this sample, but newer scales have been developed since this trial and should be used in future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT03906240/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT03906240/SAP_001.pdf
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT03906240/ICF_002.pdf